CLINICAL TRIAL: NCT02616874
Title: An Open Label Phase I Trial to Evaluate the Safety and Effect of HIVconsv Vaccines in Combination With Histone Deacetylase Inhibitor Romidepsin on the Viral Rebound Kinetic After Treatment Interruption in Early Treated HIV-1 Infected Individuals (BCN02-Romi)
Brief Title: Study to Evaluate the Safety and Effect of HIVconsv Vaccines in Combination With Histone Deacetylase Inhibitor Romidepsin on the Viral Rebound Kinetic After Treatment Interruption in Early Treated HIV-1 Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IrsiCaixa (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other); Hospital Clinic of Barcelona (Other); Hospital de Sant Pau (Other); HIVACAT (Unknown); University of Oxford (Other); BCN Checkpoint (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCN02-Romi
Record Dates: First submitted 2015-11-09; First posted 2015-11-30 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HIV
Keywords: HIV infection; Early treatment; Romidepsin; HDACi; Therapeutic Vaccines; HIVconsv; HIV reservoir; Population PK/PD analysis
MeSH Terms: conditions — HIV Infections | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MVA.HIVconsv plus romidepsin (Experimental): MVA.HIVconsv plus romidepsin
  Interventions: Drug: MVA.HIVconsv vaccine; Drug: Romidepsin

INTERVENTIONS:
Drug: MVA.HIVconsv vaccine — Dose: 2x10e8 pfu, Interval: weeks 0 and 9.
Drug: Romidepsin — Dose: 5mg/m2 over 4hours, Interval: weeks 3, 4 and 5

SUMMARY:
The BCN02-Romi study aims to evaluate a combined "kick and kill" strategy using the most immunogenic candidate vaccine available so far (HIVconsv) with the strongest latency reversal agent available at present time (romidepsin) in a cohort of early-treated HIV positive individuals.

DETAILED DESCRIPTION:
The combined use of therapeutic vaccination and specific drugs that can reactivate latent virus from the reservoir (Kick and kill strategies) hold the promise to achieve functional cure and viral eradication of HIV infection. The present project consists of a proof-of-concept clinical trial in a cohort of 24 early treated HIV-1 infected individuals rolled-over from the BCN01 vaccine clinical trial in which participants received the most immunogenic vaccines tested to date, ChAd and modified vaccinia Ankara (MVA).HIVconsv vaccines. All individuals will be given a booster immunization with MVA.HIVconsv in combination with romidepsin (RMD), a potent histone deacetylation inhibitor (HDACi) and will later undergo a monitored antiretroviral pause. HIVconsv vaccines have specifically been designed to stimulate a broad and potent cytotoxic T cell (CTL) response towards the most conserved viral regions of the HIV-1 proteome, which have recently been suggested to have a crucial role when targeting HIV variants harboured in the latent reservoir with mutations to escape T-cell immune responses. The study includes the development of a population pharmacokinetic/pharmacodynamic (PK/PD) substudy to analyse the in vivo effects of RMD in the induction of HIV expression in resting cells, deeply investigate any unintended effect on the CTL function as well as predict the relationship between RMD exposure and such effects. The investigators' results will allow investigators to optimize RMD dosing, to evaluate the clinical efficacy of this eradication strategy after the cART interruption and to identify better correlates of control of rebound viremia after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject included in ChAd-MVA.HIVconsv_BCN01 study with complete follow-up and included in BCN01-RO extension study.
2. Optimal virological suppression for at least 3 years.cop/ml).
3. Being on a non-boosted integrase-inhibitor based regimen (raltegravir or dolutegravir) for at least 4 weeks at screening visit.
4. Haematological and biochemical laboratory parameters as follows:

   * Haemoglobin > 10g/dl
   * Platelets > 100.000/dl
   * Alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
   * Creatinine ≤ 1.3 x ULN
5. CD4 T cell count ≥500 cells/mm3

Exclusion Criteria:

1. Positive pregnancy test.
2. Presence of resistance drug mutations in the screening genotype
3. History of autoimmune disease other than HIV-related auto-immune disease.
4. Treatment for cancer or lymphoproliferative disease within 1 year of study entry
5. Any other prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study
6. Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with grade >=3 adverse events assessed by Division of AIDS (DAIDS) grading table | Through study completion, maximum 75 weeks
  Grade >=3 adverse events
Number of participants with serious adverse events | Through study completion, maximum 75 weeks
  Serious adverse events
Viral reservoir measured by total HIV-1 DNA copies per 10e6 CD4+ T cells | From baseline to visit week 6 (romidepsin 3 + 1 week)
  Total HIV-1 DNA copies per 10e6 CD4+ T cells

SECONDARY OUTCOMES:
Romidepsin Cmax | week 3
  RMD plasma concentrations will be measured by Liquid chromatography-mass spectrometry (LC-MS/MS)
Romidepsin Cmax | week 4
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin Cmax | week 5
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin Cmin | week 3
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin Cmin | week 4
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin Cmin | week 5
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin area under curve (AUC) | week 3
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin AUC | week 4
  RMD plasma concentrations will be measured by LC-MS/MS
Romidepsin AUC | week 5
  RMD plasma concentrations will be measured by LC-MS/MS
HIV-1 expression in resting CD4+ T-cells measured by CA-RNA and single-copy assay (SCA) | week 6
Levels of Histone H3 acetylation in lymphocytes | week 6
CTL toxicity assessment based on viability, activation or exhaustion (most relevant marker according to previous studies) | week 6
HIVconsv-specific T cell responses will be measured by IFNg ELISPOT using peptide pools covering different HIV proteins and HIVcons sequences. | week 6
Viral suppressive capacity of CD8+ T cells in vitro, using a flow cytometric assay | Baseline
Viral suppressive capacity of CD8+ T cells in vitro, using a flow cytometric assay | Week 17
Proportion of individuals who initiate a MAP following the futility analysis | Week 17
Proportion of individuals who maintain sustained plasma viral load (pVL) <2,000 copies/ml | Week 29
Proportion of individuals in whom cART is reinitiated due to viral rebound | Up to 51 weeks
Emergence of viral resistance during MAP phase | Up to 51 weeks
  Description of viral resistance emerged, genotype.
Proportion of patients with viral suppression 6 months after treatment resumption. | 24 weeks after treatment resumption (up to 75 weeks).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Clinic Hospital, Barcelona

REFERENCES:
- [Derived] Munoz-Moreno JA, Carrillo-Molina S, Martinez-Zalacain I, Miranda C, Manzardo C, Coll P, Meulbroek M, Hanke T, Garolera M, Miro JM, Brander C, Clotet B, Soriano-Mas C, Molto J, Mothe B; BCN02-Neuro Substudy Group. Preserved central nervous system functioning after use of romidepsin as a latency-reversing agent in an HIV cure strategy. AIDS. 2022 Mar 1;36(3):363-372. doi: 10.1097/QAD.0000000000003121. PMID 34750296